CLINICAL TRIAL: NCT03942575
Title: The Risk of Postoperative Wound Complications Following the Use of Avelle Negative Pressure Wound Therapy in Patients Undergoing Mastectomy and Flap fiXation: a Pilot Study
Brief Title: The Risk of Postoperative Wound Complications Following the Use of Negative Pressure Wound Therapy in Patients Undergoing Mastectomy
Acronym: ALEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, James van Bastelaar, Surgeon, Principal Investigator, MD, PhD, Zuyderland Medisch Centrum
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METCZ20190024
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Wound Complication; Wound Infection; Wound Dehiscence; Wound Necrosis
Keywords: Negative pressure wound therapy
MeSH Terms: conditions — Breast Neoplasms; Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: A prospective cohort will be compared to a historical control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No negative pressure wound therapy (No Intervention): Historical cohort: patients who underwent mastectomy with flap fixation using tissue glue and sutures and closed suction drainage and where negative wound pressure therapy has been omitted
- Negative pressure wound therapy (Experimental): Prospective cohort: patients who underwent mastectomy with flap fixation using tissue glue and sutures and closed suction drainage with negative wound pressure therapy
  Interventions: Device: Negative pressure wound therapy

INTERVENTIONS:
Device: Negative pressure wound therapy — Wound dressing with negative pressure on closed incisions
  Arms: Negative pressure wound therapy

SUMMARY:
To evaluate the risk of postoperative wound complications following the use of Avelle negative pressure wound therapy in patients undergoing mastectomy and flap fixation, which might serve as a basis for a randomized controlled trial

DETAILED DESCRIPTION:
Rationale:

Patients and breast cancer surgeons are frequently confronted with complications after mastectomy. These complications are manifold and mainly consist of: surgical site infections, seroma, wound dehiscence and wound necrosis. These complications are caused by numerous variables and therefore a multifactorial approach is required. Due to extensive research over the years, insight has been gained in how to reduce the rate of surgical site infections and wound healing problems. For example, pre-operatively and intra-operatively the complication rate can partly be influenced by optimizing intrinsic patient factors before surgery and using prophylactic antibiotics (1). There is however room for improvement in the postoperative phase. Negative pressure wound therapy (NPWT) has proven to be useful in reducing wound complications in all sorts of wounds. Limited evidence has been published on NPWT after breast cancer surgery and the effect of such in reducing wound complications.

This is a pilot study to evaluate the effect of negative pressure wound therapy in reducing postoperative wound complications after mastectomy, which might serve as a basis for a randomized controlled trial..

Objective:

To evaluate the risk of postoperative wound complications following the use of Avelle negative pressure wound therapy in patients undergoing mastectomy and flap fixation, which might serve as a basis for a randomized controlled trial

Study design:

A prospective cohort will be compared to a historical control group. Fifty consecutive patients will undergo mastectomy with flap fixation using tissue glue and skin sutures, closed suction drainage AND Avelle negative pressure wound therapy.

These results will be compared to the results of a historical control group consisting of 112 patients who have undergone mastectomy with flap fixation using tissue glue and sutures and closed suction drainage and in whom negative wound pressure therapy was omitted.

Follow-up will be conducted for three months post mastectomy.

Study population:

Female patients > 18 years diagnosed with invasive breast cancer or DCIS ( ductal carcinoma in situ) with an indication to perform mastectomy.

Intervention (if applicable):

Application of Avelle negative pressure wound therapy after standard mastectomy with flap fixation and closed suction drainage.

Main study parameters/endpoints:

Patients with postoperative wound complications during the first three postoperative months.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients will be informed about the study before inclusion in the outpatient clinic. Informed consent will be obtained in the outpatient clinic a week after patients were initially informed. Postoperative check-ups will be done more frequently. Standard postoperative check-ups are planned at one week and three months. Additional study postoperative check-up will be performed at six weeks. Therefore, patients will be required to undergo one additional check-up. During out patients' visits, wound complication will be evaluated. Application of Avelle negative pressure wound therapy is expected to reduce wound complications and thereby benefit the post mastectomy wound healing process. The only potential risk for the patient is that the wound therapy would be ineffective or that the patient could develop an allergic reaction to the product. The latter is also a known risk of standard wound dressings.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Female sex
* Indication for mastectomy or modified radical mastectomy

Exclusion Criteria:

* Patients undergoing breast conserving therapy
* Patients undergoing direct breast reconstruction
* Unable to comprehend implications and extent of study and sign for informed consent
* Participation in other study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with post-operative wound complications | During the first three postoperative months
  Number of patients with post-operative wound complications defined as follows:
  1. Surgical site infection (SSI) is defined as redness, pain, heat or swelling at the site of the incision or by the drainage of pus. Infection rate will be measured by A) the need for antibiotics, B) seroma aspiration due to infection or C) surgical drainage during the first three postoperative months.
  2. Wound necrosis. Defined as a wound with necrotic tissue that consists of an accumulation of dead cells, tissue and cellular debris and often requires debridement.
  3. Wound dehiscence or breakdown defined as a wound that ruptures along a surgical incision and the edges of the wound no longer align.

SECONDARY OUTCOMES:
Number of unplanned visits to the ER or breast cancer clinic | During the first three postoperative months
  Number of unplanned visits to the ER or breast cancer clinic. Planned visits are standard follow-up outpatient clinic visits which are defined preoperatively. Unplanned visits are defined as any visit to the outpatient clinic which is necessary due to an adverse event.
Number of patients with clinically significant seroma | During the first three postoperative months
  Number of patients with clinically significant seroma. This is defined as:
  1. Wound healing is at risk due to seroma (wound break down, seroma leakage, necrosis)
  2. There is discomfort or pain caused by large amounts of seroma, characterised by tenseness of the skin.
  3. There is contaminated/ infected seroma and aspiration is necessary to treat infection. All patients that undergo seroma aspiration due to infection will also be treated with a one week course of Augmentin 625 mg 3 times daily.

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medisch Centrum, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Rooij L, van Kuijk SMJ, van Haaren ERM, Janssen A, Vissers YLJ, Beets GL, van Bastelaar J. Negative pressure wound therapy does not decrease postoperative wound complications in patients undergoing mastectomy and flap fixation. Sci Rep. 2021 May 5;11(1):9620. doi: 10.1038/s41598-021-89036-3. PMID 33953312